CLINICAL TRIAL: NCT03464370
Title: Evaluation of Stress Sensitivity and Hyperemotivity in Temporal Lobe Epilepsy With Enlarged Amygdala Compared to Epilepsy Without Enlarged Amygdala (Temporal and Extra-temporal) and a Group of Healthy Volunteers: Pilot Study.
Brief Title: Evaluation of Stress Sensitivity and Hyperemotivity in Epilepsy Compared to and a Group of Healthy Volunteers
Acronym: STELLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0276; 2017-A02853-50 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy
Keywords: amygdala enlargement; temporal lobe epilepsy; stress; attentional bias; anxiety; depression; PTSD
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This pilot study is prospective, monocentric, epidemiologic, case control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TLE-AE Group (Experimental): 30 subjects Age between 18 and 65 case-control with 2 witnesses per sex and age matched cases (within 5 years) for the evaluation of the primary endpoint. For the secondary endpoints, 3 controls will be matched for each case on gender and age (within 5 years) Measure of emotional stressors then evaluate the traumatic events and to date them with respect to the beginning of epilepsy in different populations of epileptics.
  Interventions: Other: Measure of emotional stressors
- Non AE epileptic Group (Active Comparator): 30 subjects Age between 18 and 65 case-control with 2 witnesses per sex and age matched cases (within 5 years) for the evaluation of the primary endpoint. For the secondary endpoints, 3 controls will be matched for each case on gender and age (within 5 years) Measure of emotional stressors then evaluate the traumatic events and to date them with respect to the beginning of epilepsy in different populations of epileptics.
  Interventions: Other: Measure of emotional stressors
- Extra-temporal epilepsy Group (Active Comparator): 30 subjects Age between 18 and 65 case-control with 2 witnesses per sex and age matched cases (within 5 years) for the evaluation of the primary endpoint. For the secondary endpoints, 3 controls will be matched for each case on gender and age (within 5 years) Measure of emotional stressors and then evaluate the traumatic events and to date them with respect to the beginning of epilepsy in different populations of epileptics.
  Interventions: Other: Measure of emotional stressors
- Healthy volunteers Group (Active Comparator): 30 subjects Age between 18 and 65 case-control with 2 witnesses per sex and age matched cases (within 5 years) for the evaluation of the primary endpoint. For the secondary endpoints, 3 controls will be matched for each case on gender and age (within 5 years) Measure of emotional stressors
  Interventions: Other: Measure of emotional stressors

INTERVENTIONS:
Other: Measure of emotional stressors — For the Epileptic Group
  * Rapid interrogation, completing the clinical data
  * A scale of impact of the precipitating factors of crises
  * An emotional Stroop
  * A task of detecting emotional targets against threatening information
  * A measure of the perception of emotions using film clips
  * A scale of measurement of perceived stress
  * The transfer of psychiatric scales
  For the healthy volunteers group :
  * A rapid interrogation, gathering the possible medical history, the level of studies, the manual laterality
  * An emotional Stroop
  * A task of detecting emotional targets against threatening information
  * A scale of measurement of perceived stress
  * A measure of the perception of emotions using film clips
  * A rapid neuropsychological assessment

SUMMARY:
Recently, a possible subtype of temporal lobe epilepsy (TLE) has been proposed: this subtype presents ipsilateral amygdala enlargement (AE) without any other lesion. However, little is known about its clinical and psychiatric phenotype. The amygdala seems to play a major role in stress related disorders (including perception of stress). The hypothesis in this study is that patients with TLE-AE more frequently report emotional distress as a seizure-precipitating factor than any other epileptic patient.

DETAILED DESCRIPTION:
TLE-AE could concern 16 to 64 % of the TLE with "negative" MRI (Beh et al., 2016).

TLE-AE patients may suffer from anxiety and depression (Lv et al, 2014). In clinical practice, it has been also identified an emotional vulnerability in these patients, as they report more frequently a high sensitivity to emotional distress than other epileptic patients. They also report a change in their affect intensity or a hyperemotivity, which appeared at the onset of their epilepsy. Lanteaume et al. have linked some TLE with an increased emotional vulnerability (Emo-TLE): these TLE patients reported stress factors precipitating their seizures. They found that the Emo-TLE group was characterized by an attentional bias toward threatening stimuli versus neutral stimuli, and that this bias was noticed neither in the TLE group without emotional vulnerability nor in healthy volunteers. But they did not study amygdala structure in each group.In the large database of the Toulouse University Hospital, screening was done to retrospectively collect TLE patients with AE identified on MRI. This large database has served to establish a reading grid in order to help the visual identification of an AE.The investigators propose to these patients them a series of validated scales to test:

* The impact of emotional stress factors for precipitating seizures
* The perception of stress (PSS-10).
* Psychiatric comorbidities (anxiety, depression, post-traumatic stress disorder, emotional lability…).

The study also propose cognitive tasks to search for an attentional bias towards threatening stimuli (Emotional Stroop and modified probe test). After this, the study will assess their emotional subjective responses (valence, arousal, avoidance) through a task during which they are presented with short movies that elicit six different emotions. At the same time, the measure of the variations of their neurovegetative system in terms of blood pressure, heart rate variability and electrodermal skin conductance variability will be done.

For each TLE-AE patient, additional healthy controls will be matched (2 for testing the primary outcome, 3 for the secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

- For all epileptic patients: Age between 18 and 65. Epilepsy (TLE or not) followed by an epileptologist.

- For TLE-AE: An AE identified on the MRI by an expert neuroradiologist. MRI must be less than one year.

- For non AE epileptic patients: No AE reported in the MRI by an expert neuroradiologist.

Exclusion Criteria:

* Any mental disorder.
* Any diabetes
* Beta-blockers
* Neuroleptics
* Any neurologic diseases for the healthy volunteers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Score on the scale of emotional seizure precipitant the outbreak | 30 minutes
  It is a hetero-questionnaire, subjectively measuring the sensitivity of an epileptic patient to the stressors of daily life that may trigger or promote the onset of their seizures.

SECONDARY OUTCOMES:
Score of The Emotional Stroop tasks | 30 minutes
  The score of the congruency index in the Emotional Stroop tasks : evaluate the attention bias towards threatening information
Score of The congruency index | 30 minutes
  The score of the congruency index in the modified probe detection tasks : evaluate the attention bias towards threatening information
Score of the Scale measures during the movie tasks | 30 minutes
  The score of scale (valence, arousal, avoidance) in the movie tasks : evaluate the emotional experience using film clips inducing emotion
Score of The Perceived Stress Scale 10 | 30 minutes
  The score of the Perceived Stress Scale 10 : evaluate the perception of stress
Score of The Tyrer's brief Scale for Anxiety (BAS) | 30 minutes
  The score of the Tyrer's brief Scale for Anxiety (BAS) will evaluate the existence of an anxiety syndrome.This scale is validated, it is a hetero-questionnaire to evaluate anxiety, in 10 items, sides from 0 to 6.
Score of The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E). | 30 minutes
  The score of the Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) : the existence of a depressive syndrome.
Score of The Affect intensity measure (AIM) | 30 minutes
  The score of the Affect intensity measure (AIM) : the multidimensional assessment of thymic states (MAThyS) : evaluate the emotional lability
Score of The Clinical-administered PTSD Scale (CAPS) | 30 minutes
  The clinical post-traumatic stress disorder scale (CAPS: Clinical-administered PTSD Scale) is the gold standard for diagnosing Post-Traumatic Stress Disorder (PTSD). To pass the entire questionnaire, it takes about sixty minutes. For the scoring list of milestones, it takes about 5 minutes. The CAPS is the only questionnaire that provides information on both the frequency and intensity of symptoms, with specific behavioral anchor points.
Score of The Post-Traumatic Checklist Scale (PCLS). | 30 minutes
  The Post-Traumatic Checklist Scale (PCLS) is a simple self-questionnaire of about 10 minutes measuring the three main sub-syndromes of post-traumatic stress disorder: repetition (items 1 to 5), avoidance ( items 6 to 12) and neurovegetative hyperactivity (items 13 to 17). The scale is composed of 17 items, rated from 1 to 5. There is a cut-off at ≥ 45 to diagnose post-traumatic stress disorder. The validity of the French translation has been verified.

CONTACTS AND LOCATIONS:
Overall Officials: Marie DENUELLE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No